

| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Version Number: | 3.1 |
| | Effective Date: | 25-Nov-2021 |

## Statistical Analysis Plan

## **Study Title**

A prospective, multi-centre, phase IV clinical trial to assess the safety and efficacy of Acalabrutinib capsules in Indian adult Patients with chronic lymphocytic leukaemia and relapsed and refractory mantle cell lymphoma

| Protocol/ Study Number | : | D8220C00022 | |
|---|---|---|---|
| Sponsor Name | : | AstraZeneca Pharma India Limited | |
| Sponsor Addre s | : | AstraZeneca Pharma India Limited | |
| | | Block N1, 12th Floor, Manyata Embassy | |
| - X | | Business Park | |
| | | Rachenahalli, Outer Ring Road, | |
| | ), | Bangalore-560045 | |
| Document Version | : 🕊 | 1.0 | |
| Document Date | : | 17-Jan-2022 | |
| | | 44 | |
| Author Name (s) : | : | PPD | |
| Designation | : | Biostatistician | |
| | | | 500 |
| | | Cy | |
| | | | 20 |
| | | | 44 |
| | | | $\sim$ |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# **Table of Contents**

| LIST OF TABLE | 4 |
|--------------------------------------------------------|--------------|
| LIST OF LISTING | 5 |
| LIST OF FIGURES | 5 |
| LIST OF ABBREVIATION | 7 |
| 1. INTRODUCTION | 8 |
| 2. Study Objective and Design | 8 |
| 2.1 Study Objective | 8 |
| 2.1.1 Primary Objective | 8 |
| 2.1.2 Secondary Objective | 8 |
| 2.2 Study Description | 8 |
| 2.2.1 Study Design | 8 |
| 2.2.2 Inclusion Criteria | 9 |
| 2.2.3 Exclusion Criteria | 11 |
| 2.2.4 Study Flow Chart | 12 |
| 2.2.5 Study Plan | 13 |
| 2.3 Randomization | 15 |
| 2.4 Blinding and Un-Blinding | 15 |
| 2.5 Interim Analysis | 15 |
| 3. Population Analysis Set | 15 |
| 3.1 Full Analysis Set | 15 |
| 4. Sample Size and Power Calculations | 16 |
| 5. Patient Characteristics and Study Conduct Summaries | 16 |
| 5.1 General Considerations | 16 |
| 5.2 Decimal Point | 16 |
| 5.3 Disposition of Patients | 16 |
| 5.4 Demographic and Baseline Characteristics | 16 |
| 6. Efficacy Analysis Strategy | 17 |
| 6.1 Efficacy Endpoints | 17 |
| 6.1.1 Primary Endpoint | 17 |
| 6.1.2 Secondary Endpoint | 17 |
| 6.2 Efficacy Hypothesis | 17 |
| 6.3 Statistical Methods for Efficacy Analysis | 17 |
| Document | Page 2 of 72 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| 6.3.1 Primary Endpoint Analysis | 17 |
|-----------------------------------|----|
| 6.3.2 Secondary Endpoint Analysis | 18 |
| 7. References | 18 |
| 8. Mock Tables | 19 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## LIST OF TABLE

| Table 14.1.1. Patient Disposition in the Study | 19 |
|-------------------------------------------------------------------|-----|
| Table 14.1.2. Summary of Demographic and Baseline Characteristics | 20 |
| Table 14.1.3. Summary of Medical and Surgical History | 21 |
| Table 14.1.4. Summary of Concomitant Medication | 22 |
| Table 14.1.5. Summary of Baseline Disease Characteristics | 23 |
| Table 14.1.6. Summary of Lymph Node Biopsy | 24 |
| Table 14.1.7. Summary of Next Generation Sequencing-CLL | 25 |
| Table 14.1.8. Summary of Chest X-Ray | 26 |
| Table 14.1.9. Summary of urine Pregnancy Test | 27 |
| Table 14.2.1. Analysis of Objective Response | 28 |
| Table 14.2.2. Summary of QLQ-C30 Questionnaire | 29 |
| Table 14.3.1. Summary of Adverse Event | 333 |
| Table 14.3.2. Summary of Physical examination | 34 |
| Table 14.3.3. Summary of Electrocardiogram | 35 |
| Table 14.3.4.1. Summary of Laboratory assessment for Haematology | 36 |
| Table 14.3.4.2. Summary of Laboratory assessment for Biochemistry | 37 |
| Table 14.3.4.3. Summary of Laboratory assessment for Serology | 38 |
| Table 14.3.5. Summary of Vital Signs | 39 |
| Table 14.3.6. Summary of ECOG | 40 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## LIST OF LISTING

| Listing 16.2.1.1. Listing of Patient Informed Consent Details | 41 |
|----------------------------------------------------------------------|----|
| Listing 16.2.1.2. Listing of Patient Study Completion | 42 |
| Listing 16.2.2. Listing of Patient Demographics | 43 |
| Listing 16.2.3. Listing of Patient Baseline Disease characteristics | 44 |
| Listing 16.2.4. Listing of Patient Lymph Node Biopsy | 45 |
| Listing 16.2.5. Listing of Patient Next Generation Sequencing-CLL | 46 |
| Listing 16.2.6. Listing of Patient Medical or Surgical History | 47 |
| Listing 16.2.7.1. Listing of Patient Acalabrutinib dosing (Part I) | 48 |
| Listing 16.2.7.2. Listing of Patient Acalabrutinib dosing (Part II) | 49 |
| Listing 16.2.7.3. Listing of Patient Treatment Compliance | 50 |
| Listing 16.2.8. Listing of Patient Chest X-ray | 51 |
| Listing 16.2.9.1. Listing of Patient CT Scan and MRI | 52 |
| Listing 16.2.9.2. Listing of Patient Response Assessment | 53 |
| Listing 16.2.10. Listing of Patient QLP-C30 Questionnaire | 54 |
| Listing 16.2.11.1. Listing of Patient Adverse event log (Part I) | 57 |
| Listing 16.2.11.2. Listing of Patient Adverse event log (Part II) | 58 |
| Listing 16.2.12.1. Listing of Patient SAE (Part I) | 59 |
| Listing 16.2.12.2. Listing of Patient SAE (Part II) | 60 |
| Listing 16.2.13. Listing of Patient Physical Examination | 61 |
| Listing 16.2.14. Listing of Patient ECG Performed. | 62 |
| Listing 16.2.15.1. Listing of Patient Haematology | 63 |
| Listing 16.2.15.2. Listing of Patient Biochemistry | 64 |
| Listing 16.2.15.3. Listing of Patient Urinalysis | 65 |
| Listing 16.2.15.4. Listing of Patient Serology | 66 |
| Listing 16.2.16. Listing of Patient Vital Signs | 67 |
| Listing 16.2.17. Listing of Patient ECOG | 68 |
| Listing 16.2.18.1. Listing of Patient Urine Pregnancy test | 69 |
| Listing 16.2.18.2. Listing of Patient Pregnancy From | 70 |
| Listing 16.2.19. Listing of Patient Concomitant Medications | 71 |
| Listing 16.2.20. Listing of Patient Prior and Concomitant medication | 72 |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## LIST OF FIGURES

Not Applicable



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## LIST OF ABBREVIATION

| AE | Adverse Event |
|---|---|
| AESI | AEs of special interest |
| ALT | Alanine Aminotransferase |
| ANC | Absolute Neutrophil Count |
| BID | Twice daily |
| BTK | Bruton Tyrosine Kinase |
| CLL | Chronic Lymphocytic Leukaemia |
| CMV | Cytomegalovirus |
| CNS | Central Nervous System |
| CR | Complete Remission |
| СТ | Computed Tomography |
| CTCAE | Common Terminology Criteria for Adverse Event |
| ECG | Electrocardiography |
| ECOG | Eastern Cooperative Oncology Group |
| EORTC QLQC30 | European Organization for the Research and Treatment of Cancer |
| | Quality of Life Questionnaire |
| Hb | Haemoglobin |
| HCV | Hepatitis C Virus |
| HIV | Human Immunodeficiency Virus |
| ICH | International Conference on Harmonisation |
| IGHV | Immunoglobulin Variable Heavy Chain |
| iwCLL | International Workshop on Chronic Lymphocytic Leukaemia |
| LDT | Lymphocyte Doubling Time |
| MCL | Mantle Cell Lymphoma |
| MedDRA | Medical Dictionary for Regulatory Activities |
| MRI | Magnetic Resonance Imaging |
| PI | Prescribing Information |
| PR | Partial Remission |
| PRL | Partial Response with Treatment-Induced Lymphocytosis |
| PRO | Patients-reported outcome |
| SAE | Serious Adverse Event |
| SLL | Small Lymphocytic Lymphoma |
| SoA | Schedule of Activities |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## 1. INTRODUCTION

The purpose of this document is to provide a description of the statistical methods and procedures to be implemented for the analysis of data from D8220C00022 study. This document is based on protocol version 1.0 Dated 01-SEP-2020. The statistical planning and conduct of analysis of the data from this study will follow the principles defined in relevant ICH-E9 guidelines. Any change from the planned analysis as described in the protocol, are detailed here, and any differences described here supersede the analysis as presented in the protocol.

## 2. Study Objective and Design

## 2.1 Study Objective

## 2.1.1 Primary Objective

 To investigate the safety of Acalabrutinib among Patients with treatment naïve and R/R CLL/ SLL, and relapsed & refractory MCL in Indian Patient

#### 2.1.2 Secondary Objective

- To assess the efficacy of Acalabrutinib in Patients of CLL/SLL and relapsed & refractory MCL in Indian Patients.
- Patient-reported outcome (PRO)

## 2.2 Study Description

## 2.2.1 Study Design

The study is a phase IV, open-label, single-arm, multi-centre, prospective study to be conducted in India. The study will evaluate the safety and efficacy of Acalabrutinib in Indian adult Patients with CLL/SLL and Patients with MCL who have received at least one prior therapy. The Investigator will be trained on the locally approved Prescribing Information (PI) before the enrolment of the first Patient at their site to ensure compliance and proper dosing of the study drug. Patients will be monitored throughout the study period for AEs /SAEs/AESI of Acalabrutinib.

Patients with CLL/SLL and MCL who are eligible to receive Acalabrutinib treatment as per locally approved PI and ratified by an independent clinical judgment of treating physician will be evaluated for inclusion into the current phase IV trial. To enrol approximately 100 Patients (90 Patients of TN & R/R CLL and 10 R/R MCL Patients) into the study, it is expected that approximately 150 Patients will need to be screened.

The study will be initiated after approval by the Ethics Committee. Patients will undergo the following phases: Screening/Enrolment Phase, Treatment Phase, and Follow-up Phase.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

The decision of Patients to participate in this study must not, in any way, impact the standard of care they are receiving or any benefits to which they are otherwise entitled. Prior to data collection, all Patients must sign an Informed Consent Form (ICF), allowing for data collection and source data verification to be performed in accordance with local requirements and Sponsor policy.

Two cohorts of Patients will be included in the current study (a) Patients with CLL/SLL who are treatment naïve or have received at least one prior therapy (N= 90) and (b) Patients with MCL who have received at least one prior therapy (N= 10). Potential Patients will undergo screening phase within 07 days prior to the first dose. Patients who meet the protocol-defined inclusion/exclusion criteria will be prospectively enrolled in the study. Acalabrutinib capsules 100 mg are administered twice daily (BID) for 06 cycles, starting from Cycle 1, Day 1, and continuing up to Cycle 6, Day 28; or until study drug discontinuation due to either disease progression or, unacceptable toxicity, or other reasons, whichever occurs earlier.

Acalabrutinib will be provided by the Sponsor to Patients in the Treatment Phase. The Sponsor shall also conduct laboratory investigations for safety and efficacy evaluations, including haematology, biochemistry, radiology, and electrocardiography (ECG), as mentioned in the SoA table.

## 2.2.2 Inclusion Criteria

- 1. Men and Women aged 18yrs or more.
- 2. Eastern Cooperative Oncology Group (ECOG) performance status of 0,1, or 2
- 3. Able to receive all outPatient treatments, all laboratory monitoring, and all radiologic evaluations.
- 4. The following laboratory parameters:
  - a. Absolute neutrophil count (ANC) ≥750 cells/μL or ≥500 cells/μL in Patients with documented bone marrow involvement, and independent of growth factor support 07 days before the assessment
  - b. Platelet count ≥50,000 cells/μL or ≥30,000 cells/μL in Patients with documented bone marrow involvement, and without transfusion support 07 days before the assessment
  - c. Aspartate transaminase (AST) and Alanine transaminase (ALT) ≤2.0 x ULN
  - d. Total bilirubin ≤1.5 x ULN
  - e. Estimated creatinine clearance of ≥30 mL/min
- 5. Refractory disease defined as achieving less than partial response with the most recent treatment within 6 months before study entry
- 6. Provision of signed, written and dated informed consent prior to any study-specific Procedures
- 7. The Patients of either CLL or MCL:
  - a. CLL Patients:



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

- i. Treatment naïve or ≥1 prior systemic therapy for CLL
- ii. Diagnosis of CD20+ CLL that meets published diagnostic criteria (Hallek et al. 2018)
- iii. An active disease that meets ≥1 of the following iwCLL 2018 criteria for requiring treatment:
  - 1) Evidence of progressive marrow failure as manifested by the development of, or worsening of, anaemia and/or thrombocytopenia. Cut-off levels of Hb <10 g/dL or platelet counts <100 × 109/L are generally regarded as an indication for treatment. However, in some Patients, platelet counts <100 × 109/L may remain stable over a long period; this situation does not automatically require therapeutic intervention.</p>
  - 2) Massive (i.e., ≥6 cm below the left costal margin) or progressive or symptomatic splenomegaly.
  - Massive nodes (i.e., ≥10 cm in longest diameter) or progressive or symptomatic lymphadenopathy.
  - 4) Progressive lymphocytosis with an increase of ≥50% over a 2-month period or Lymphocyte Doubling Time (LDT) in <6 months. LDT can be obtained by linear regression extrapolation of absolute lymphocyte counts obtained at intervals of 2 weeks over an observation period of 2 to 3 months; Patients with initial blood lymphocyte counts <30 × 109/L may require a longer observation period to determine the LDT. Factors contributing to lymphocytosis other than CLL (e.g., infections, steroid administration) should be excluded.</p>
  - Autoimmune complications, including anaemia or thrombocytopenia poorly responsive to corticosteroids.
  - 6) Symptomatic or functional extra-nodal involvement (e.g., skin, kidney, lung, spine).
  - 7) Disease-related symptoms as defined by any of the following:
    - a) Unintentional weight loss of ≥10% within the previous 06 months.
    - b) Significant fatigue (i.e., ECOG performance scale 02 or worse; cannot work or unable to perform usual activities).
    - c) Fever ≥100.5°F or 38.0°C for 02 or more weeks without evidence of infection.
    - d) Night sweats for ≥1 month without evidence of infection.

#### b. MCL Patients:

- i. Confirmed MCL with translocation t(11;14) (q13;q32) and/or overexpressed cyclin D1
- ii. Measurable nodal disease (one or more lesions measuring ≥2 cm in the longest diameter)
- iii. Relapsed after, or were refractory to, 1-5 previous treatments.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

#### 2.2.3 Exclusion Criteria

- 1. Known prolymphocytic leukaemia, Central Nervous System (CNS) lymphoma or leukaemia; or known history of (or currently suspected) Richter's syndrome
- 2. Treatment with chemotherapy, external beam radiation therapy, anticancer antibodies, or investigational drug within 30 days of the first dose of study drug
- 3. Prior radio-conjugated or toxin-conjugated antibody therapy
- 4. Anticoagulation therapy (e.g., warfarin or equivalent vitamin K antagonists) within 07 days of the first dose of study drug.
- 5. Major surgery ≤30 days before the first dose of study drug
- 6. History of stroke or intracranial haemorrhage ≤6 months before the first dose of study drug.
- 7. History of bleeding diathesis
- 8. Prior exposure to a B-cell lymphoma-2 (Bcl-2) inhibitor or B-cell receptor inhibitor like BTKs
- Active Cytomegalovirus (CMV) infection or serologic status reflecting active Hepatitis B or C infection or known history of infection with Human Immunodeficiency Virus (HIV), or any uncontrolled active systemic infection.
- 10. Significant cardiovascular disease such as uncontrolled or symptomatic arrhythmias, Congestive Heart Failure, or Myocardial Infarction within 06 months of screening, or any Class 3 or 4 cardiac diseases as defined by the New York Heart Association Functional Classification, or QTcB >480 msec at screening.
- 11. Requiring treatment with proton-pump inhibitors (e.g., Omeprazole, Esomeprazole, Lansoprazole, Dexlansoprazole, Rabeprazole, or Pantoprazole).
- 12. Breastfeeding or pregnant.
- 13. Current life-threatening illness, medical condition, or organ/system dysfunction which, in the Investigator's opinion, could have compromised the Patient's safety or put the study at risk.
- 14. Concurrent participation in another therapeutic clinical trial.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## 2.2.4 Study Flow Chart





| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## 2.2.5 Study Plan

| Study Phase | Screening<br>Phase | Treatment Phase * | | Follow-up<br>Phase |
|---|---|---|---|---|
| Cycle | 1 | Cycles 1-6 | EOT | EOS |
| Visit No. | 1 | 2-7 (Day 1 of each cycle) | 8 | |
| Study Days | -6 to 0 | 1-168 (28 days per<br>cycle) | 170 | 28 days post-<br>EOT |
| Screening/Enrolment visit | | | | 100 |
| Informed consent 8 | X | | | |
| Eligibility Criteria | x | 1 | | |
| Demographics/ Review<br>medical history | x | | | |
| ECOG Performance Status | X | X | X | |
| General Physical<br>examination <sup>b</sup> | X | Symptom-directed physical examination only | | |
| Concomitant medication recording | THE R. P. LEWIS CO., LANSING, MICH. 499, 187, 197, 197, 197, 197, 197, 197, 197, 19 | from the time of ICF<br>ib dose in the treatment pl | And the second of the second o | after the last |
| Study Drug Administration | | | | |
| Acalabrutinib dosing | | The recommended dose<br>100 mg capsules BID, s<br>Cycle 1, until disease<br>unacceptable toxicity.<br>treatment is 28 days. | starting on Day 1<br>progression or | |
| Disease Evaluations (Disease | characteristics | will be performed as per | routine clinical p | ractice) |
| Baseline Disease<br>Characteristics | x | | | |
| Safety Evaluations (baseline | and each treatn | nent visit) * | t. | • |
| Physical examination <sup>b</sup> | X | Symptom-directed physexamination only | sical | |
| Vital parameters ° | X | X | X | Ü |
| Adverse event monitoring | | ontinuous from the time of ICF until 28 days after last study dose of calabrutinib. | | |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Study Phase | Screening<br>Phase | Treatment Phase * | | Follow-up<br>Phase |
|---|---|---|---|---|
| Cycle | | Cycles 1-6 | EOT | EOS |
| Visit No. | 1 | 2-7 (Day 1 of each cycle) | 8 | |
| Study Days | -6 to 0 | 1-168 (28 days per<br>cycle) | 170 | 28 days post-<br>EOT |
| 12-lead ECG | х | X | X | |
| Lymph node biopsy <sup>d</sup> | x | | | |
| Next-generation<br>sequencing (NGS)-CLL<br>panel <sup>c</sup> | x | | | |
| Haematology <sup>f</sup> &<br>Biochemistry <sup>g</sup> | x | х | x | 1 |
| Urinalysis h | X | X | X | |
| Pregnancy Test i | x | x | X | |
| Chest X-ray i | X | x | X | |
| Efficacy Evaluations (once i | n 3 months) | | • | • |
| CT/MRI k | x | X | X | |
| EORTC QLQ-C30<br>Questionnaire | x | х | x | |

<sup>\$</sup> Patients must sign the informed consent form before any study-specific procedures are performed.

- a. Treatment phase from Day 1 to Day 168. The treatment with Acalabrutinib will be continued until disease progression or unacceptable drug-related toxicity, whichever occurs earlier.
- b. The screening physical examination will include, at a minimum, the general appearance of the Patient, height (screening only) and weight, and examination of the skin, eyes, ears, nose, throat, lungs, heart, abdomen, extremities, musculoskeletal system, lymphatic system, and nervous system. Symptomdirected physical examination, including tumour assessments by palpation, are done thereafter.
- c. Vital signs (blood pressure, heart rate, and temperature) will be assessed after the Patient has rested in the sitting position.

<sup>\*</sup> Procedures conducted as part of the Patient's routine clinical management (e.g., blood count) and obtained before signing of the Informed Consent Form (ICF) may be utilised for screening or baseline purposes provided the procedures meet the protocol-specified criteria and were performed within the time frame (-6 to 0 day)



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

d. Lymph node biopsy will be conducted in Patients with lymphadenopathy. However, a report of previous lymph node biopsy performed within 06 months before the study enrolment could be considered if the Patient did not receive any medication during that period

| Study Phase | Screening<br>Phase | Treatment Phase <sup>a</sup> | | Follow-up<br>Phase |
|---|---|---|---|---|
| Cycle | | Cycles 1-6 | EOT | EOS |
| Visit No. | 1 | 2-7 (Day 1 of each cycle) | 8 | |
| Study Days | -6 to 0 | 1-168 (28 days per cycle) | 170 | 28 days post-<br>EOT |

- e. Next-generation sequencing will be conducted to understand the genetic profile in Indian settings. Molecular cytogenetics (FISH) for del(13q), del(11q), del(17p), trisomy 12 in peripheral blood lymphocytes; TP53 mutation; immunoglobulin variable heavy chain (IGHV) mutational status will be assessed before the start of treatment in CLL/SLL-naïve Patients, or CLL/SLL Patients who did not have their report. However, MCL Patients are Relapsed/Refractory and their previous report data will be used. A six months old report can be considered for both the conditions.
- f. Haematology will include a complete blood cell count [white blood cell count, haemoglobin (Hb), haematocrit, reticulocyte, and platelet count] and differential leukocyte count, including both percent and an absolute number of lymphocytes. Haematology need not be repeated on Cycle 1 Day 1 if screening haematology was within 5 days.

#### 2.3 Randomization

Not Applicable

## 2.4 Blinding and Un-Blinding

Not Applicable

## 2.5 Interim Analysis

Interim analyses is planned for first 50 subjects who completes the study. All the primary safety analysis will be produced for the interim analysis.

## 3. Population Analysis Set

## 3.1 Full Analysis Set

The Full Analysis Set (FAS) will consist of all enrolled Patients who received at least one dose of Acalabrutinib.

| Proprietar | v and | Confid | lentia | l Document |
|------------|-------|--------|--------|------------|
|------------|-------|--------|--------|------------|



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

The FAS will be used for all analyses of safety and efficacy.

## 4. Sample Size and Power Calculations

The primary endpoint of the trial is to demonstrate the safety profile of Acalabrutinib in routine clinical practice as assessed by the incidence of adverse events (AEs) (Serious and Non-serious AEs) observed during the trial. As per the Health Authority requirement, the total sample size of the study will be approximately 100.

## 5. Patient Characteristics and Study Conduct Summaries

#### 5.1 General Considerations

Statistical Analysis will be performed using SAS (version 9.4 or higher) software (SAS Institute Inc USA). Categorical variables will be summarized with the frequency and percentage of Patients in each category. Continuous variables will be summarized descriptively with the number of Patients, mean, standard deviation, minimum, median and maximum values.

#### 5.2 Decimal Point

Unless otherwise noted, means, median, will be presented to one decimal place more than the measured value, the same decimal as the measured value, percentages and confidence intervals will be presented to two decimal places and p-value will be presented to three decimal place. Percentages after zero counts will not be displayed and percentages equating to 100% will be presented as 100%, without any decimal places.

#### 5.3 Disposition of Patients

Patient disposition table will be based on all enrolled Patients who consented to participate in the study. The following summaries will be included in the disposition table: total number of Patients screened in the study, number and percentage of Patients who failed screening, number and percentage of Patients who completed the study, and number and percentage of Patients who discontinued from the study with reason for discontinuation.

## 5.4 Demographic and Baseline Characteristics

Demographic and baseline characteristics will be summarized based on the Full Analysis Set.

Descriptive summaries will be provided for the demographic and baseline characteristics. Demographic characteristics and baseline characteristics such as Age, Gender, Height, Race, etc. will be summarized and tabulated for Full Anlyssis set.

All the continuous variables (i.e., age, height etc.) will be summarized by n, mean, standard deviation, minimum, median and maximum values. All the categorical variables will be summarized as counts and percentages.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Chatishical Analysis Blan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## 6. Efficacy Analysis Strategy

## 6.1 Efficacy Endpoints

## 6.1.1 Primary Endpoint

 Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESI) including Arrhythmias (Atrial Fibrillation), Anaemia, Hypertension, Bleeding, Infections, Reasons for discontinuation and second primary malignancies

### 6.1.2 Secondary Endpoint

- Objective response to treatment.
- Health related quality of life (EORTC QLQC30 Questionnaire)

### 6.2 Efficacy Hypothesis

#### Not Applicable

## 6.3 Statistical Methods for Efficacy Analysis

All primary and secondary efficacy endpoints will be summarized by Full Analysis Set.

Categorical data will be summarized using frequencies and percentages. Continuous data will be summarized with descriptive statistics, including mean, standard deviation, median, minimum, and maximum.

## 6.3.1 Primary Endpoint Analysis

Primary Endpoint evaluations will include adverse event monitoring, physical examinations, ECG monitoring, clinical laboratory investigations (haematology and biochemistry), vital sign measurements, ECOG performance status and death as observed by the Investigator.

Adverse Events (AEs), Serious Adverse Events (SAEs), and AEs of Special Interest (AESI) will be summarized using frequencies and percentages.

Physical examination will be collected as per visit scheduled. Physical examination results (normal /abnormal) from scheduled visits will be summarized for each body system. A listing will be provided for the Normal/abnormal physical examination parameters.

A 12-lead electrocardiogram (ECG) will be performed as per visit scheduled. ECG results (normal, abnormal clinically insignificant, abnormal clinically significant) will be summarized as counts and percentage.

Laboratory investigations (haematology and biochemistry) data will be collected as per visit scheduled. Laboratory values will be presented using the International System of Units (SI units). Observed values will be summarized descriptively (n, mean, median, standard deviation, minimum, and maximum values). A listing will be provided which contains data for each laboratory parameter.



| | Document Title: | Document ID: | BP04-01 |
|---|---|---|---|
| | Chalishing Angloris Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 | |

Vital signs will be performed as per visit scheduled. Vital signs parameters include Systolic Blood Pressure, Diastolic Blood Pressure, Heart Rate, Respiratory rate and Temperature. Descriptive summaries (n, mean, median, standard deviation, minimum and maximum values) of observed values in each vital sign parameter at each assessment visit will be presented. A listing will be provided for all vital signs parameters assessments.

ECOG will be performed as per visit scheduled. ECOG performance status will be summarized as counts and ercentage.

### 6.3.2 Secondary Endpoint Analysis

Secondary Endpoint evaluations will be assessed based on iwCLL 2018 criteria for CLL/SLL and for MCL. Efficacy will be based on objective response [Complete Remission (CR) + Partial Remission (PR) and Partial response with lymphocytosis (PRL)] via Computed Tomography (CT) scans or Magnetic Resonance Imaging (MRI). The sum of complete response and partial responses and Partial response with lymphocytosis (PRL)] will be summarized using frequencies, percentage and 95% CI will be calculated using Clopper Pearson confidence interval method. Health related quality of life (EORTC QLQC30 Questionnaire) summarized using frequencies and percentage.

## 7. References

- D8220C00022 Protocol, Version No: 01, AstraZeneca Pharma India Limited, Block N1, 12th Floor, Manyata
   Embassy, Business Park, Rachenahalli, Outer Ring Road, Bangalore-560045
- ICH E3 Guideline
- ICH E9; STATISTICAL PRINCIPLES FOR CLINICAL TRIALS.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## 8. Mock Tables

Table 14.1.1. Patient Disposition in the Study

| | CLL/SLL<br>(N=xx) | MCL<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| Patients Screened | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Screen Failures | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Patients Completed the study | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Patients Discontinued the study | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Reason for Discontinuation | | | |
| Patient Decision | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Adverse Event | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Severe non-compliance to study protocol | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Initiation of alternative anticancer therapy including another investigational agent | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Disease progression | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Pregnancy or intent to become pregnant | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Other | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Other 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Other 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number of all Enrolled Patients.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Patients Screened", "Screen Failures", "Patient completed the study" and "Patients Dicontinued the study" rows are based on the number of Patient in each group.
- Percentages in the "Reasons for Discontinuation" rows are based on the number of Patients Discontinued study in each group.
- Note: Screened Patients are those who signed the informed consent
- Source :Listing 16.2.1.1, listing 16.2.1.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.2. Summary of Demographic and Baseline Characteristics

| | CLL/SLL | MCL | Total |
|---|---|---|---|
| Demographic and Baseline Variables | (N=xx) | (N=xx) | (N=xx) |
| Age (Years) | | | |
| n | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Gender | | | |
| Male | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Female | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Missing | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Race | | | |
| Asian | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Other | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Other 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Other n | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Height (cm) | | | |
| n | xx | XX | xx |
| Missing | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages are based on number of patient in each group.
- SD = Standard Deviation, min=minimum, max=maximum
- Source :Listing 16.2.2.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Applysis Plan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.3. Summary of Medical and Surgical History

| System Organ Class / Preferred | CLL/SLL | MCL | Total |
|----------------------------------|------------|------------|------------|
| Term | (N=xx) | (N=xx) | (N=xx) |
| | n (%) | n (%) | n (%) |
| Patient with any medical history | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| System Organ Class 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| System Organ Class 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| System Organ Class 3 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| System Organ Class 4 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| System Organ Class 5 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Preferred Term 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Patient with any medical history" rows are based on number of patient in each group.
- Percentages in the "System Organ Class" and "Preferred Term" rows are based on number of Patient with any medical history in each group.
- Medical histories were coded using MedDRA Ver23.0
- Source :Listing 16.2.6



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Dlan | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.4. Summary of Concomitant Medication

| | CLL/SLL<br>(N=xx) | MCL<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|
| <del>-</del> | n (%) | n (%) | n (%) |
| Visit 1 | 11 (70) | 11 (76) | 11 (70) |
| Any concomitant medication given during visit | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Any prior therapy received for Chronic Lymphocytic | , , | . , | |
| Leukemia/ Mantle Cell Lymphoma | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Patient refractory to the Therapy | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Visit x | | | |
| Any New Concomitant medication given Since Last | | | |
| Visit | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages are based on number of patient in each group.
- Programme Note: Visit x- Visit 2 up to Visit 8.
- Source :Listing 16.2.19



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.5. Summary of Baseline Disease Characteristics

| | CLL/SLL | MCL | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| | n (%) | n (%) | n (%) |
| Clinical Staging (Rai Staging) of Chronic Lymphocytic | | | |
| Leukaemia | | , , | |
| Stage 0 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage I | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage II | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage III | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage IV | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Characteristics | | | |
| Only Blood abnormality | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Blood abnormality with lymphadenopathy | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Blood abnormality with organomegaly | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| CLL-IPI Score | | | |
| n | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Mantle Cell Lymphoma | | | |
| Relapsed | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Refractory | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Clinical Staging (Ann Arber) | | | |
| Stage I | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage II | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage IE | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage IIE | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage III | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage IIIS | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage IIIE | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Stage IV | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Genomic alteration | | | |
| Translocation t(11;14) (q13;q32) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Overexpressed cyclin D1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| MIPI Score | . , | . , | . , |
| n | XX | xx | xx |
| Missing | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages are based on number of patient in each group.
- SD = Standard Deviation, min=minimum, max=maximum
- Source :Listing 16.2.3.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.6. Summary of Lymph Node Biopsy

| | CLL/SLL | MCL | Total<br>(N=xx) |
|---|---|---|---|
| | (N=xx) | (N=xx) | |
| | n (%) | n (%) | n (%) |
| Lymph node enlarged | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Size of Lymph node (mm) | | | |
| n | XX | XX | XX |
| Missing | XX | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Lymph node biopsy performed within 6 months before study enrolment | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Method of Biopsy | | | |
| Fine-needle aspiration biopsy | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Core needle biopsy | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Open (surgical) biopsy | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages are based on number of patient in each group.
- SD = Standard Deviation, min=minimum, max=maximum
- Source :Listing 16.2.4.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.1.7. Summary of Next Generation Sequencing\_CLL

| | (N=xx) |
|-----------------------------------------------------------|------------|
| | n (%) |
| Genomic sample collected for molecular cytogenetics (FISH | 1) |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| NA | xx (xx.xx) |
| Any genomic alteration observed | |
| Yes | xx (xx.xx) |
| No | xx (xx.xx) |
| If Yes | |
| 11q deletion | xx (xx.xx) |
| 13q deletion | xx (xx.xx) |
| 17p deletion | xx (xx.xx) |
| 12 addition | xx (xx.xx) |
| TP53 mutation | xx (xx.xx) |
| IGHV mutation | xx (xx.xx) |
| Other | xx (xx.xx) |
| Other 1 | xx (xx.xx) |
| Other n | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Genomic sample collected for molecular cytogenetics" and "Any Genomic alteration observed" rows are based on number of patient in each group.
- Percentages in the "If yes" rows are based on number of Patient Any genomic alteration observed.
- Source :Listing 16.2.5.



| Document Title: | Document ID: | BP04-01 |
|-----------------|--------------|---------|
| Effective Date: | 25-Nov-2021 | |

Table 14.1.8. Summary of Chest X-Ray

| | CLL/SLL | MCL | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| _ | n (%) | n (%) | n (%) |
| Visit x | | | |
| Patient have any sign and symptom of Pneumonia | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Views | | | |
| Posteroranterior | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Anteroposterior | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Lateral | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Assessment Result | | | |
| Normal | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Abnormal | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| If abnormal | | | |
| Unilateral | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Bilateral | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| If Unilateral | | | |
| Unilobar | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Bilobar | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentage in the "Patient have any Sign and Symptoms of Pneumonia" rows are based on number of patient in each group
- Percentage in the "Views" rows are based on the Number of Patient have any Sign and Symptoms of Pneumonia in each group.
- Programmer Note Visit x: Visit 1 up to Visit 8
- Source :Listing 16.2.8.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.1.9. Summary of urine Pregnancy Test

| | CLL/SLL | MCL<br>(N=xx)<br>n (%) | Total<br>(N=xx)<br>n (%) |
|---|---|---|---|
| | (N=xx) | | |
| | n (%) | | |
| Visit x | | | |
| Urine Pregnancy Test Performed | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Result | | | |
| Positive | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Negative | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Programmer Note Visit x: Visit 1 up to Visit 8.
- Percentage in the "Urine Pregnanacy Test" row based on number of patient in each group.
- Percentages in the "Result" row are based on the number of Patient with urine Pregnancy Test performed in each group.
- Source :Listing 16.2.18.1



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Table 14.2.1. Analysis of Objective Response

| | CLL/SLL | MCL | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| | n (%) | n (%) | n (%) |
| Visit 5 | | | |
| Response Assessment | | | |
| Complete Response (CR) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Partial Response (PR) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Partial Response with lymphocytosis (PR-L) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Objective response | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 95 % CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |
| Visit 8 | • • • | , , , | |
| Response Assessment | | | |
| Complete Response (CR) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Partial Response (PR) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Partial Response with lymphocytosis (PR-L) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Objective response | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 95 % CI | (xx.x, xx.x) | (xx.x, xx.x) | (xx.x, xx.x) |

- Objective response =Complete Response (CR) + Partial Response (PR) + Partial Response with lymphocytosis (PRL)
- Percentage in the "Reponse Assessment" are based on number of patient in each group.
- 95 % CI will be calculated based on clopper Pearson confidence interval method
- Source :Listing 16.2.9.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.2.2. Summary of QLQ-C30 Questionnaire

| | CLL/SLL<br>(N=xx) | MCL<br>(N=xx) | MCL<br>(N=xx) |
|---|---|---|---|
| • | n (%) | n (%) | n (%) |
| Visit x | , , | ` , | |
| Do you have any trouble doing strenuous activities, like carrying a heavy | | | |
| shopping bag or a suitcase | | | |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Do you have any trouble taking a long walk | , , | | |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Do you have any trouble taking a short walk outside of the house | , | , | , , |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Do you need to stay in bed or a chair during the day | ^^ (^^.^^) | ** (*****) | ~~ (~~.~~) |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | | | |
| · | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Do you need help with eating, dressing, washing yourself or using the toilet | | | |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | xx (xx.xx)<br>xx (xx.xx) | | |
| | | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Were you limited in doing either your work or other daily activities | ( | / | ( |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Were you limited in pursuing your hobbies or other leisure time activities | | | |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Were you short of breath | | | |
| 1 (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Have you had pain | , , | , , | , , |
| | | D | 20 -6 72 |
| Document | | rage | 29 of 72 |



| | Document Title: | Document ID: | BP04-01 | |
|---|---|---|---|---|
| | | Version Number: | 3.1 | |
| | Statistical Analysis Plan | Effective Date: | 25-Nov-2021 | |
| ١ | | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Dic | d you need to rest | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| На | ve you had trouble sleeping | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| На | ve you felt weak | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| На | ve you lacked appetite | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| На | ve you felt nauseated | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| На | ve you vomited | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| На | ve you been constipated | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| На | ve you had diarrhea | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| We | ere you tired | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Γ | Document | | Раде | 30 of 72 |
| L | p era j ana communition populition | | . 450 | |



| | Document Title: | Document ID: | BP04-01 | |
|---|---|---|---|---|
| | Charterian Amakada Dian | Version Number: | 3.1 | |
| | Statistical Analysis Plan | Effective Date: | 25-Nov-2021 | |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Die | d pain interfere with your daily activities | | | |
| | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | ve you had difficulty in concentrating on things, like reading | | , | , , |
| | wspaper or watching television | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | d you feel tense | ( | (, | , |
| | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | d you worry | ^^ (^^.^^) | ^^ (^^.^^) | ^^ (^^.^^) |
| | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Quite a bit) | | xx (xx.xx)<br>xx (xx.xx) | xx (xx.xx)<br>xx (xx.xx) |
| | | xx (xx.xx) | | |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | d you feel irritable | and an and | var (var var) | , a., (, a., , a., ) |
| | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | d you feel depressed | | , , | , , |
| | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | ve you had difficulty remembering things | | | |
| | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | s your physical condition or medical treatment interfered ware<br>nily life | ith your | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | (Quite a bit) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (Very much) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | s your physical condition or medical treatment interfered w | | , , | . , |
| | cial activities | | | |
| 1 | (Not at all) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| | (A little) | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| [ | Document | | Page | 31 of 72 |



| | Document Title: | Document ID: | BP04-01 | |
|---|---|---|---|---|
| | Statistical Analysis Plan Version Nu Effective D | | 3.1 | |
| \$ | | | 25-Nov-2021 | |
| 3 (Quite a bit) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Has your physical co | ndition or medical treatment caused you | financial | | |
| difficulties | | | | |
| 1 (Not at all) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 (A little) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 (Quite a bit) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 (Very much) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| How would you rate | your overall health during the past week | | | |
| 1 (Very Poor ) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 5 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 6 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 7 (Excellent) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| low would you rate | your overall quality of life during the pas | t week | | |
| 1 (Very Poor ) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 5 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 6 | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 7 (Excellent) | | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| otal Score | | | | |
| n | | XX | xx | XX |
| Missing | | XX | XX | XX |
| Mean (SD) | | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx |
| Median | | XX.X | XX.X | XX.X |
| (min, max) | | (xx.xx, xx.xx | ) (xx.xx, xx.xx) | (xx.xx, xx.x |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Programmer Note Visit x: Visit 1, Visit 5 and Visit 8
- Percentage are based on number of patient in each group.
- Source :Listing 16.2.10.



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.1. Summary of Adverse Event

| | CLL/SLL | MCL | Total |
|---|---|---|---|
| | (N=xx) | (N=xx) | (N=xx) |
| | n (%) | n (%) | n (%) |
| Patient Experience Any Adverse Event | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| CTCAE grade | | | |
| Mild | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Moderate | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Severe | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Life – Threatening or disabling | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Death | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Investigator's causality rating against the Investigational Pro | oduct | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Action Taken | | | |
| None | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Non-drug treatment required | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Hospitalization/ prolonged hospitalization | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Diagnostic or clinical test(s) conducted | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Drug Withdrawn | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Patient Withdrawn | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Treatment taken | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Outcome | | | |
| Recovered without sequelae | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Recovered with sequelae | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Not recovered/ Not resolved | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Recovering/ resolving | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Unknown | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Fatal | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Patient Experience Any Adverse Event" rows are based on number of patient in each group.
- Percentages in the "CTCAE grade, Investigator's causality rating against the Investigational Product, Action Taken,
   Patient Withdrawn, Treatment taken and Outcome" rows are based on number of Patient Experience Any Adverse Event in each group.
- Source :Listing 16.2.11.1, Listing 16.2.11.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.2. Summary of Physical examination

| | CLL/SLL<br>(N=xx) | MCL<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|
| | n (%) | n (%) | n (%) |
| Visit x | | | |
| Physical examination performed | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| System x | | | |
| Normal | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Abnormal NCS | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Abnormal CS | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentages in the "Physical Examination performed" rows are based on number of patient in each group.
- Percentages in the "System x" rows are based on number of Patient Physical Examination performed in each group.
- Programmer Note: Generate summaries for the following System x: General Appearance, Skin, Eyes, Ears, Nose, Throat, Lungs, Heart, Abdomen, Extermities, Musculoskeletal System, Lymphatic System, Nervous System, Liver, Spleen and Other.
- NCS= Non-clinically significant
- CS= clinically significant
- Programme Note: Visit x- Visit 1 up to Visit 8
- Source :Listing 16.2.13



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.3. Summary of Electrocardiogram

| | CLL/SLL<br>(N=xx) | MCL<br>(N=xx) | Total<br>(N=xx) |
|------------------|-------------------|----------------|-----------------|
| Visit x | (** ****) | (** ****) | (12.11.4) |
| ECG Performed | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Heart rate (bpm) | , , | , , | , , |
| n | xx | XX | XX |
| Missing | xx | xx | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| QRS (ms) | , | , , , | , , , |
| n | xx | XX | XX |
| Missing | xx | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | xx.x | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| PR (ms) | , | , | , |
| n | xx | XX | xx |
| Missing | xx | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| RR (ms) | | | |
| n | xx | XX | xx |
| Missing | xx | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| QT (ms) | | | |
| n | xx | XX | xx |
| Missing | xx | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| QTcB (ms) | • | | |
| n | xx | XX | xx |
| Missing | xx | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum
- Visit x: Visit 1 up to Visit 8
- Source :Listing 16.2.14



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.4.1. Summary of Laboratory assessment for Haematology

| | CLL/SLL<br>(N=xx) | MCL<br>(N=xx) | Total<br>(N=xx) |
|---|---|---|---|
| Visit x | | | |
| Sample Collected | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Haematology Parameter x | | | |
| n | Xx | Xx | Xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum
- Percentages in the "Sample collected" rows are based on number of patient in each group.
- Programmer Note: Generate summaries for the following Haematology parameters x: Haematocrit (%), Haemoglobin (g/dL), Neutrophils (%), Basophils (%), Eosinophils (%), Monocytes(%), Absolute Lymphocytes Count(thou/μL), Percentage Lymphocytes (%), Reticulocyte (%), Absolute Neutrophils Count (thou/μL), Platelet Count (thou/μL), Total leukocyte count(thou/μL).
- Programmer Note Visit x: Visit 1 up to Visit 8
- Source :Listing 16.2.15.1


| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.4.2. Summary of Laboratory assessment for Biochemistry

| | CLL/SLL | MCL | Total |
|--------------------------|----------------|----------------|----------------|
| | (N=xx) | (N=xx) | (N=xx) |
| Visit x | | | |
| Sample Collected | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Biochemistry Parameter x | | | |
| n | xx | XX | XX |
| Missing | xx | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum
- Percentages in the "Sample collected" rows are based on number of patient in each group.
- Programmer Note: Generate summaries for the following parameters x Albumin (g/dL), Glucose (mg/dL), Amylase (U/L), Lipase (U/L), Alkaline phosphatase (U/L), Lactate dehydrogenase (U/L), Alanine aminotransferase (U/L), Aspartate aminotransferase (U/L), Potassium (mmol/L), Bicarbonate (mmol/L), Sodium (mmol/L), Calcium (mg/dL), Total bilirubin (mg/dL), Chloride(mmol/L), Total Protein (g/dL), Creatinine (mL/min/1.73m²), Urea (mg/dL), Blood Urea Nitrogen (mg/dL), Gamma-glutamyltransferase (U/L), Magnesium (mg/dL), Haptoglobin (g/L) and b2-microglobulin(ng/ML).
- Programmer Note Visit x: Visit 1 up to Visit 8.
- Source :Listing 16.2.15.2



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.4.3. Summary of Laboratory assessment for Serology

| | CLL/SLL<br>(N=xx) | MCL | Total<br>(N=xx) |
|---|---|---|---|
| | | (N=xx) | |
| | n (%) | n (%) | n (%) |
| Sample Collected | | | |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| HIV | | | |
| Positive | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Negative | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Active Cytomegalovirus (CMV) infection | | | |
| Positive | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Negative | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Hepatitis B surface antigen (HBsAg) | | | |
| Positive | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Negative | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Hepatitis B surface antibody (HBsAb) | | | |
| Positive | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Negative | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Anti-HBc antibody | | | |
| Positive | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Negative | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Anti-HCV antibody | | | |
| Positive | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Negative | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentage rows are based on number of patient in each group
  Percentage in the "HIV", "Active Cytomegalovirus (CMV) infection"," Hepatitis B surface antigen (HBsAg)"," Hepatitis B surface antibody (HBsAb)"," Anti-HBc antibody" and "Anti-HCV antibody" rows are based on /nuber of Patient Sample Collected.
- Source :Listing 16.2.15.4



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Table 14.3.5. Summary of Vital Signs

| | CLL/SLL | MCL<br>(N=) | Total |
|---|---|---|---|
| Mil-to | (N=xx) | (N=xx) | (N=xx) |
| Visit x | | | |
| Vital Signs Collected | , , | , , | , , |
| Yes | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| No | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| Weight (Kg) | | | |
| n | Xx | Xx | Xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | XX.X | XX.X | XX.X |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Heart rate (bpm) | | | |
| n | Xx | Xx | Xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Respiratory rate (Breaths/min) | | | |
| n | Xx | Xx | Xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | XX.X | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Systolic Blood Pressure (mmHg) | | | |
| n | Xx | Xx | Xx |
| Missing | Xx | Xx | Xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Diastolic Blood Pressure (mmHg) | , , , | , , , | , , , |
| n | xx | xx | xx |
| Missing | xx | XX | XX |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | xx.x | xx.x | xx.x |
| (min, max) | (xx.xx, xx.xx) | (xx.xx, xx.xx) | (xx.xx, xx.xx) |
| Temperature (F) | (Animy Anim) | (Many Many | (runny runny |
| n | XX | xx | xx |
| Missing | XX | XX | xx |
| Mean (SD) | xx.x (xx.xx) | xx.x (xx.xx) | xx.x (xx.xx) |
| Median | | | |
| (min, max) | xx.x<br>(xx.xx, xx.xx) | xx.x<br>(xx.xx, xx.xx) | xx.x<br>(xx.xx, xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- SD = Standard Deviation, min=minimum, max=maximum ;Percentage rows are based on the number of Full Analysis Set.
- Visit x: Visit 1 up to Visit 8; Source: Listing 16.2.16



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

### Table 14.3.6. Summary of ECOG

| ECOG performed | CLL/SLL<br>(N=xx) | MCL<br>(N=xx) | Total<br>(N=xx) |
|----------------|-------------------|---------------|-----------------|
| • | n (%) | n (%) | n (%) |
| Visit x | | | |
| ECOG Grade | | | |
| 0 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 1 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 2 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 3 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 4 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |
| 5 | xx (xx.xx) | xx (xx.xx) | xx (xx.xx) |

- The Capital "N" in the column header represents the total number Full Analysis Set.
- The small "n" in summary statistics represents the total number of Patients.
- Percentage rows are based on number of patient in each group.
- Programme Note: Visit x- Visit 1 up to Visit 8.
- Source :Listing 16.2.17



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

# Listing 16.2.1.1. Listing of Patient Informed Consent Details

| Patient Number | Patient Group | Informed consent | Date and Time for Informed Consent |
|---|---|---|---|
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY/HH:MM |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.2.1.2. Listing of Patient Study Completion

| Patient | | Patient completed | Date of study | Primary reason | |
|---|---|---|---|---|---|
| Number | Patient Group | the study | completion/discontinuation | for withdrawal | Other, specify |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | Xxxx | Xxxx |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XXXX | XXXX |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XXXX | XXXX |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XXXX | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.2. Listing of Patient Demographics

| Patient Number | Patient Group | Age/Gender | Date of Birth | Height (cm) | Race | Other, Specify |
|---|---|---|---|---|---|---|
| xx-xxxx | (CLL/SLL)/(MCL) | xx/xxx | DD-MMM-YYYY | xxx | XXXX | XXXX |
| XX-XXXX | (CLL/SLL)/(MCL) | xx/xxx | DD-MMM-YYYY | XXX | XXXX | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.3. Listing of Patient Baseline Disease characteristics

| Patient | | Date of | Clinical Staging of Chronic | | CLL-IPI | Mantle Cell | | Genomic | MIPI |
|---|---|---|---|---|---|---|---|---|---|
| Number | Patient Group | Diagnosis | Lymphocytic Leukaemia | Characteristics | Score | Lymphoma | Clinical Staging | Alteration | Score |
| XX-XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | xx | XXXX | xxxx | Relapsed / Refractory | XXXX | xxxx | xxxx |
| XX-XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | xx | XXXX | xxxx | Relapsed / Refractory | XXXX | xxxx | xxxx |
| XX-XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | xx | XXXX | xxxx | Relapsed / Refractory | XXXX | xxxx | xxxx |
| XX-XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | xx | XXXX | XXXX | Relapsed / Refractory | XXXX | xxxx | xxxx |
| XX-XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | XX | XXXX | XXXX | Relapsed / Refractory | XXXX | XXXX | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.4. Listing of Patient Lymph Node Biopsy

| | | lymp | Lymp | lymph node | lymph node biopsy performed Patient receive any medication | | | |
|---|---|---|---|---|---|---|---|---|
| <b>Patient</b> | | node | node | biopsy | within 6 | | for the study indication from | Method |
| Number | Patient Group | enlarged | (mm) | required | months before study enrolment | Date of biopsy | day of biopsy till date | of Biopsy |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | Yes/No | Yes/No | DD-MMM-YYYY | Yes/No | Xxxx |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | Yes/No | Yes/No | DD-MMM-YYYY | Yes/No | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.2.5. Listing of Patient Next Generation Sequencing-CLL

| Patient<br>Number | Genomic sample collected for molecular cytogenetics (FISH) | Date of sample | Any genomic alteration observed | Specify the alterations | Other,<br>specify |
|---|---|---|---|---|---|
| XX-XXXX | Yes/No/NA | DD-MMM-YYYY | Yes/No | xxxx | xxxx |
| XX-XXXX | Yes/No/NA | DD-MMM-YYYY | Yes/No | XXXX | xxxx |
| XX-XXXX | Yes/No/NA | DD-MMM-YYYY | Yes/No | XXXX | xxxx |
| XX-XXXX | Yes/No/NA | DD-MMM-YYYY | Yes/No | xxxx | XXXX |
| XX-XXXX | Yes/No/NA | DD-MMM-YYYY | Yes/No | XXXX | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.6. Listing of Patient Medical or Surgical History

| Patient | | Patient have any medical | Seq. | Medical/Surgical | System | Preferred | | | | Received |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Patient Group | or Surgical History | No | History Description | Organ Class | Term | Start Date | Stop Date | Ongoing | Treatment |
| xx-xxxx | (CLL/SLL)/(MCL) | Yes/No | XX | XXXX | XXXX | xxxx | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | Yes/No |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No | XX | XXXX | XXXX | XXXX | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.7.1. Listing of Patient Acalabrutinib dosing (Part I)

| Patient | | | Capsule Acalabrutinib | Number of Capsule | IP kit | Acalabrutinib |
|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | dispensed for cycle 1 | dispensed | Number | administered at the visit |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XX | XXXXXX | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.2.7.2. Listing of Patient Acalabrutinib dosing (Part II)

| | | | Capsule | Capsule | Capsule | Capsule | Capsule | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| | | | Acalabrutinib | Acalabrutinib | Acalabrutinib | Acalabrutinib | Acalabrutinib | Number of | | Acalabrutinib |
| <b>Patient</b> | | | dispensed for | dispensed for | dispensed for | dispensed for | dispensed for | Capsule | IP kit | administered |
| Number | Visit | Patient Group | cycle 2 | cycle 3 | cycle 4 | cycle 5 | cycle 6 | dispensed | Number | at the visit |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | Yes/No | Yes/No | Yes/No | Yes/No | XX | XXXXXX | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

Listing 16.2.7.3. Listing of Patient Treatment Compliance

| Patient | | | Any change from | If Yes, | Patient 100% compliant with the treatment |
|---|---|---|---|---|---|
| Number | Visit | Patient Group | the dosing schedule | comment | medication in last treatment cycle |
| xx-xxxx | XXXX | (CLL/SLL)/(MCL) | Yes/No | Xxxx | Yes/No |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | Xxxx | Yes/No |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXXX | Yes/No |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | Xxxx | Yes/No |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | xxxx | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.2.8. Listing of Patient Chest X-ray

| Patient | | | Patient have any Sign and | | | | | If |
|---|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | Symptom of Pneumonia | Date and Time for Image | Views | Assessment Result | If abnormal | Unilateral |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY/HH:MM | XXXX | Normal/Abnormal | Unilateral/Bilateral | Unilobar/Bilobar |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.2.9.1. Listing of Patient CT Scan and MRI

| | | | CT Scan or | | | | Anteroposteri | Thick | Size of | Volume | Sum of Product | Percentage |
|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | | Patient | MRI | Date and Time | Type of | Size of spleen | or diameter | ness | the Liver | of Liver | diameter | change from |
| Number | Visit | Group | performed | for Image | Image | Length (cm) | (cm) | (cm) | (cm) | (ml) | (mm) | visit 1 (%) |
| | | (CLL/SLL)/ | | DD-MMM- | CT Scan/ | | | | | | | _ |
| XX-XXXX | XXXX | (MCL) | Yes/No | YYYY/HH:MM | MRI | XXXX | XXXX | XXXX | xxxx | XXXX | XXXX | XXXX |
| | | (CLL/SLL)/ | | DD-MMM- | CT Scan/ | | | | | | | |
| XX-XXXX | XXXX | (MCL) | Yes/No | YYYY/HH:MM | MRI | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX | XXXX |
| | | (CLL/SLL)/ | | DD-MMM- | CT Scan/ | | | | | | | |
| XX-XXXX | XXXX | (MCL) | Yes/No | YYYY/HH:MM | MRI | XXXX | XXXX | XXXX | XXXX | XXXX | Xxxx | Xxxx |
| | | (CLL/SLL)/ | | DD-MMM- | CT Scan/ | | | | | | | |
| XX-XXXX | XXXX | (MCL) | Yes/No | YYYY/HH:MM | MRI | XXXX | XXXX | XXXX | xxxx | XXXX | Xxxx | Xxxx |
| | | (CLL/SLL)/ | | DD-MMM- | CT Scan/ | | | | | | | |
| XX-XXXX | XXXX | (MCL) | Yes/No | YYYY/HH:MM | MRI | XXXX | XXXX | XXXX | XXXX | XXXX | Xxxx | Xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-----------|
| Statistical Analysis Plan | Effective Date: | nber: 3.1 |

Listing 16.2.9.2. Listing of Patient Response Assessment

| Patient Number | Visit | Patient Group | Response Assessment |
|----------------|-------|-----------------|---------------------|
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | xxxx |



| Document Title: Statistical Analysis Plan | Document ID: | BP04-01 |
|---|---|---|
| Control Andrew Dis- | Version Number: | 3.1 |
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.2.10. Listing of Patient QLP-C30 Questionnaire

| | | D -1 C | Date of | | 6 | Tota |
|---|---|---|---|---|---|---|
| Patient Number | Visit | Patient Group | Assessment | Questionnaire | Score | Scor |
| | | | | Do you have any trouble doing strenuous activities, like carrying a heavy | | |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | shopping bag or a suitcase? | XXXX | XXXX |
| | | | | Do you have any trouble taking a long walk? | XXXX | |
| | | | | Do you have any trouble taking a short walk outside of the house? | XXXX | |
| | | Do you need to stay in bed or a chair during the day? | XXXX | | | |
| | | Do you need help with eating, dressing, washing yourself or using the toilet? | XXXX | | | |
| | | | | Were you limited in doing either your work or other daily activities? | XXXX | |
| | | | | Were you limited in pursuing your hobbies or other leisure time activities? | XXXX | |
| | | Were you short of breath? | XXXX | | | |
| | | Have you had pain? | xxxx | | | |
| | | Did you need to rest? | xxxx | | | |
| | | Have you had trouble sleeping? | xxxx | | | |
| | | | | Have you felt weak? | xxxx | |
| | | | | Have you lacked appetite? | xxxx | |
| | | | | Have you felt nauseated? | xxxx | |
| | | | | Have you vomited? | xxxx | |
| | | | | Have you been constipated? | xxxx | |
| | | | | Have you had diarrhea? | xxxx | |
| | | | | Were you tired? | xxxx | |
| | | | | Did pain interfere with your daily activities? | xxxx | |
| | | | | Have you had difficulty in concentrating on things, like reading a newspaper | | |
| | | | | or watching television? | xxxx | |
| | | | | Did you feel tense? | xxxx | |
| | | | | Did you worry? | xxxx | |
| | | | | Did you feel irritable? | xxxx | |
| | | | | Did you feel depressed? | XXXX | |
| | | | | Have you had difficulty remembering things? | XXXX | |



XX-XXXX

| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| | Has your physical condition or medical treatment interfered with your family | |
|---|---|---|
| | life? | XXXX |
| | Has your physical condition or medical treatment interfered with your social activities? | 2000 |
| | | XXXX |
| | Has your physical condition or medical treatment caused you financial difficulties? | www |
| | | XXXX |
| | How would you rate your overall health during the past week? | XXXX |
| | How would you rate your overall quality of life during the past week? Do you have any trouble doing strenuous activities, like carrying a heavy | XXXX |
| DD-MMM-YYYY | , | 1000 |
| יטט-ועוועוועו-דדד | shopping bag or a suitcase? Do you have any trouble taking a long walk? | XXXX |
| | | XXXX |
| | Do you have any trouble taking a short walk outside of the house? | XXXX |
| | Do you need to stay in bed or a chair during the day? | XXXX |
| | Do you need help with eating, dressing, washing yourself or using the toilet? | XXXX |
| | Were you limited in doing either your work or other daily activities? | XXXX |
| | Were you limited in pursuing your hobbies or other leisure time activities? | XXXX |
| | Were you short of breath? | XXXX |
| | Have you had pain? | XXXX |
| | Did you need to rest? | XXXX |
| | Have you had trouble sleeping? | XXXX |
| | Have you felt weak? | XXXX |
| | Have you lacked appetite? | XXXX |
| | Have you felt nauseated? | XXXX |
| | Have you vomited? | XXXX |
| | Have you been constipated? | XXXX |
| | Have you had diarrhea? | XXXX |
| | Were you tired? | XXXX |
| | Did pain interfere with your daily activities? | XXXX |
| | Have you had difficulty in concentrating on things, like reading a newspaper | |
| | or watching television? | XXXX |
| | Did you feel tense? | XXXX |
| | Did you worry? | XXXX |

** Document** 

(CLL/SLL)/(MCL)

XXXX

Page 55 of 72

XXXX



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

| Did you feel irritable? | XXXX |
|---|---|
| Did you feel depressed? | XXXX |
| Have you had difficulty remembering things? | XXXX |
| Has your physical condition or medical treatment interfered with your family | |
| life? | XXXX |
| Has your physical condition or medical treatment interfered with your social | |
| activities? | XXXX |
| Has your physical condition or medical treatment caused you financial | |
| difficulties? | xxxx |
| How would you rate your overall health during the past week? | XXXX |
| How would you rate your overall quality of life during the past week? | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.11.1. Listing of Patient Adverse event log (Part I)

| Patient | | | Patient experience Any | Seq. | Event | System | Preferred | Start Date and Start | |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | Adverse event | No | Description | Organ Class | Term | Time | End Date and End Time |
| xx-xxxx | XXXX | (CLL/SLL)/(MCL) | Yes/No | XX | xxxx | xxxx | xxxx | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM |
| xx-xxxx | XXXX | (CLL/SLL)/(MCL) | Yes/No | XX | xxxx | xxxx | xxxx | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XX | XXXX | XXXX | XXXX | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XX | xxxx | xxxx | xxxx | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XX | XXXX | xxxx | xxxx | DD-MMM-YYYY/HH:MM | DD-MMM-YYYY/HH:MM |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.11.2. Listing of Patient Adverse event log (Part II)

| | | | | | Investigator's causality | | | | |
|---|---|---|---|---|---|---|---|---|---|
| <b>Patient</b> | | | | CTCAE | rating against the | Action | <b>Patient</b> | Treatment | |
| Number | Visit | Patient Group | Ongoing | grade | Investigational Product | Taken | Withdrawn | Taken | Outcome |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | XXXX | XXXX | Yes/No | XXXX | Yes/No | Yes/No | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | XXXX | XXXX | Yes/No | XXXX | Yes/No | Yes/No | XXXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | XXXX | XXXX | Yes/No | XXXX | Yes/No | Yes/No | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | XXXX | XXXX | Yes/No | XXXX | Yes/No | Yes/No | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | XXXX | XXXX | Yes/No | XXXX | Yes/No | Yes/No | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.12.1. Listing of Patient SAE (Part I)

| | | | | Date of Investigator | Patient | | System Organ | | |
|---|---|---|---|---|---|---|---|---|---|
| <b>Patient</b> | SAE | | Date of AE met | became aware of | Hospitalised | Date of Hospitalisation/ Date of | Class/ Preferred | Seriousness | Date of Event |
| Number | Term | Patient Group | Criteria for SAE | serious AE | due to SAE | Discharge | Term | Criteria | Onset |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY/ DD-MMM-YYYY | XXXX | XXXX | DD-MMM-YYYY |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY/ DD-MMM-YYYY | XXXX | xxxx | DD-MMM-YYYY |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY/ DD-MMM-YYYY | XXXX | XXXX | DD-MMM-YYYY |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY/ DD-MMM-YYYY | XXXX | XXXX | DD-MMM-YYYY |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | DD-MMM-YYYY | Yes/No | DD-MMM-YYYY/ DD-MMM-YYYY | XXXX | xxxx | DD-MMM-YYYY |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.12.2. Listing of Patient SAE (Part II)

| Patient | | Causality assessment in | Causality assessment in<br>relation to Other | | | Autopsy | |
|---|---|---|---|---|---|---|---|
| Number | Patient Group | relation to study procedure | medication | Outcome | Outcome Date | performed | Date of Autopsy |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No/NA | xxxx | xxxx | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No/NA | xxxx | xxxx | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No/NA | xxxx | XXXX | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No/NA | xxxx | XXXX | DD-MMM-YYYY | Xxxx | DD-MMM-YYYY |
| XX-XXXX | (CLL/SLL)/(MCL) | Yes/No/NA | xxxx | xxxx | DD-MMM-YYYY | XXXX | DD-MMM-YYYY |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.13. Listing of Patient Physical Examination

| Patient Number | Visit | Patient Group | Physical examination performed | Date of Examination | Seq. No. | System | Result |
|---|---|---|---|---|---|---|---|
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XX | XXXX | XXXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XX | xxxx | XXXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XX | xxxx | XXXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XX | XXXX | xxxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XX | XXXX | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.2.14. Listing of Patient ECG Performed.

| Patient | | | ECG | Date and Time for ECG | | | | |
|---|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | performed | performed | Parameter | Result | Unit | Finding |
| xx-xxxx | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | xxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.15.1. Listing of Patient Haematology

| Patient | | | Blood Sample | No, Specify | Date and Time for Blood | | If Other | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | collected | Reason | Sample collected | Parameter | Parameter | Result | Unit | Finding |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | xxx | DD-MMM-YYYY/HH:MM | XXX | xxx | XXX | XXX | xxx |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | XXX | XXX | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | xxx | DD-MMM-YYYY/HH:MM | XXX | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | xxx | DD-MMM-YYYY/HH:MM | XXX | xxx | XXX | XXX | xxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.15.2. Listing of Patient Biochemistry

| Patient | | | Blood Sample | No Specify | Date and Time for Blood | | If, Other | | | |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | collected | Reason | Sample collected | Parameter | Parameter | Result | Unit | Finding |
| xx-xxxx | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | xxx | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | xxx | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | xxx | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | xxx | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | xxx | DD-MMM-YYYY/HH:MM | xxx | xxx | XXX | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.15.3. Listing of Patient Urinalysis

| Patient | | | Urin Sample | No Specify | Date and Time for Urin | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | collected | Reason | Sample collected | Parameter | Result | Unit | Finding |
| xx-xxxx | XXXX | (CLL/SLL)/(MCL) | Yes/No | xxx | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | xxx | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | XXX | DD-MMM-YYYY/HH:MM | xxx | XXX | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.15.4. Listing of Patient Serology

| Patient | Blood Sample | | No Specify | Date and Time for blood | | Active Cytomegalovirus | | | Anti-HBc | Anti-HCV |
|---|---|---|---|---|---|---|---|---|---|---|
| Number | Collected | Patient Group | Reason | sample collected | HIV | (CMV) infection | HbsAg | HBsAb | antibody | antibody |
| xx-xxxx | Yes/No | (CLL/SLL)/(MCL) | Xxx | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | XXXX | xxxx |
| XX-XXXX | Yes/No | (CLL/SLL)/(MCL) | Xxx | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | xxxx | xxxx |
| XX-XXXX | Yes/No | (CLL/SLL)/(MCL) | Xxx | DD-MMM-YYYY/HH:MM | XXXX | xxxx | XXXX | XXXX | xxxx | xxxx |
| XX-XXXX | Yes/No | (CLL/SLL)/(MCL) | Xxx | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | xxxx | xxxx |
| XX-XXXX | Yes/No | (CLL/SLL)/(MCL) | Xxx | DD-MMM-YYYY/HH:MM | XXXX | XXXX | XXXX | XXXX | XXXX | xxxx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.16. Listing of Patient Vital Signs

| Patient | | | Vital Signs | Date of Vital | | | | | |
|---|---|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | Collected | Signs Collected | Parameters | Result | Unit | Finding | If, Abnormal CS |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | xxx | XXX | XXX | Xxx | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XXX | XXX | XXX | Xxx | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XXX | XXX | XXX | Xxx | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XXX | XXX | XXX | xxx | XXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | DD-MMM-YYYY | XXX | XXX | XXX | XXX | XXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

Listing 16.2.17. Listing of Patient ECOG

| Patient Number | Visit | Patient Group | Date of ECOG | ECOG Grade |
|----------------|-------|-----------------|--------------|------------|
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | Xx |
| XX-XXXX | xxxx | (CLL/SLL)/(MCL) | DD-MMM-YYYY | Xx |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.18.1. Listing of Patient Urine Pregnancy test

| Urine | | Urine Pregnancy test | No, Specify | Date and Time of | | |
|---|---|---|---|---|---|---|
| Patient Number | Visit | Patient Group | performed | Reason | Assessment | Result |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No/NA | XXX | DD-MMM-YYYY/HH:MM | Positive/Negative |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.18.2. Listing of Patient Pregnancy From

| Patient | | | Date of pregnancy | Date of last | Estimated Date of | Outcome of | If Live Birth, provide |
|---|---|---|---|---|---|---|---|
| Number | Visit | Patient Group | conformed | menstrual period | Delivery | pregnancy | the Birth Outcome |
| xx-xxxx | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | DD-MMM-YYYY | DD-MMM-YYYY | xxxx | XXXX |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | DD-MMM-YYYY | DD-MMM-YYYY | DD-MMM-YYYY | Xxxx | XXXX |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| Statistical Analysis Plan | Effective Date: | 25-Nov-2021 |

## Listing 16.2.19. Listing of Patient Concomitant Medications

| | | | Any Concomitant | Any New Concomitant | Any prior therapy received for | | Dose per | | | Patient |
|---|---|---|---|---|---|---|---|---|---|---|
| Patient | | | medication given | medication given Since | Chronic Lymphocytic | therapy | Administra | | Route of | Refractory to |
| Number | Visit | Patient Group | during Visit | Last Visit | Leukemia / Mantle Cell Lymphoma | | tion | Unit | Administration | the Therapy |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | Yes/No | Yes/No | XX | xx | Xx | XX | Yes/No |
| XX-XXXX | Xxxx | (CLL/SLL)/(MCL) | Yes/No | Yes/No | Yes/No | XX | XX | Xx | XX | Yes/No |
| XX-XXXX | Xxxx | (CLL/SLL)/(MCL) | Yes/No | Yes/No | Yes/No | XX | XX | Xx | XX | Yes/No |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | Yes/No | Yes/No | XX | XX | Xx | XX | Yes/No |
| XX-XXXX | XXXX | (CLL/SLL)/(MCL) | Yes/No | Yes/No | Yes/No | XX | xx | Xx | XX | Yes/No |



| Document Title: | Document ID: | BP04-01 |
|---------------------------|-----------------|-------------|
| | Effective Date: | 25-Nov-2021 |

## Listing 16.2.20. Listing of Patient Prior and Concomitant medication

| • | | Patient receive any | | | Preferred Term/ | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|
| Patient | Patient | prior/ concomitant | Seq. | Medication | System Organ | Start Date/ | | Indication | Dosage | Dose/ | Route/ |
| Number | Group | medications | NO | Name | Class | End Date | Ongoing | Description | Form | Unit | Frequency |
| | (CLL/SLL)/ | | | | | DD-MMM-YYYY/ | | | | xxxx/ | |
| XX-XXXX | (MCL) | Yes/No | XX | xxxx/xxxx | xxxx/xxxx | DD-MMM-YYYY | xxxx | XX | XXXX | XXXX | xxxx/xxxx |
| | (CLL/SLL)/ | | | | | DD-MMM-YYYY/ | | | | xxxx/ | |
| XX-XXXX | (MCL) | Yes/No | XX | xxxx/xxxx | xxxx/xxxx | DD-MMM-YYYY | XXXX | XX | XXXX | XXXX | xxxx/xxxx |
| | (CLL/SLL)/ | | | | | DD-MMM-YYYY/ | | | | xxxx/ | |
| XX-XXXX | (MCL) | Yes/No | XX | xxxx/xxxx | xxxx/xxxx | DD-MMM-YYYY | xxxx | XX | XXXX | XXXX | xxxx/xxxx |
| | (CLL/SLL)/ | | | | | DD-MMM-YYYY/ | | | | xxxx/ | |
| xx-xxxx | (MCL) | Yes/No | XX | xxxx/xxxx | xxxx/xxxx | DD-MMM-YYYY | xxxx | XX | XXXX | XXXX | xxxx/xxxx |
| | (CLL/SLL)/ | | | | | DD-MMM-YYYY/ | | | | xxxx/ | |
| XX-XXXX | (MCL) | Yes/No | XX | xxxx/xxxx | xxxx/xxxx | DD-MMM-YYYY | XXXX | XX | XXXX | XXXX | xxxx/xxxx |